CLINICAL TRIAL: NCT03749304
Title: Monitoring Analgesia by ANI (Analgesia The Nociception Index) During Surgery Inflammatory Bowel
Brief Title: Monitoring Analgesia by ANI (Analgesia The Nociception Index)
Acronym: ANI-MICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012_31; 2012-A01363-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Nociceptive Pain; Surgical Procedure, Unspecified
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANI monitor (Experimental)
  Interventions: Device: ANI monitor

INTERVENTIONS:
Device: ANI monitor — experimental medical device using expert rules and continuous reading of heart rate, blood pressure and Analgesia Nociception Index

SUMMARY:
The objective of this research is to study the variations of the ANI(Analgesia The Nociception Index) according to 2 periods: the "NoStim" period before surgical incision under general anesthesia and the period of hemodynamic reactivity "ReactHemo" peroperative. This period is defined by a 20% increase in FC and / or PAS (the only gold standard today).

ELIGIBILITY:
Inclusion Criteria:

* patient with IBD
* Scheduled surgery: laparotomy or laparoscopic resection with high risk of laparo-conversion

Exclusion Criteria:

* patient included in another current study or the previous month
* urgent surgery
* toxicomania or receiving opioids preoperatively
* pregnant woman
* psychosis
* betablocker treatment
* diabetic dysautonomia
* non-sinus heart rate
* pacemaker heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-03-16 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change of ANI greater than 20 points | During the surgery, an average Three hours and a half
  ANI decrease greater than 20 points between a "NoStim" period before surgical incision under general anesthesia and a period of intraoperative "ReactHemo" hemodynamic reactivity defined by a 20% increase in FC and / or PAS.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France